CLINICAL TRIAL: NCT05445349
Title: Measurement of Breathing Parameters of Asthma and COPD Patients With Different Degrees of Disease Severity for the Computer Simulation of Lung Deposition of Aerosol Drugs
Brief Title: Breathing Parameter Measurements for Lung Deposition Simulation
Acronym: CHOICE
Status: Completed | Type: Observational
Sponsor: Medisol Development Kft. (Industry)
Collaborators: Pest County Pulmonology Hospital (Unknown); University of Debrecen (Other); St. Borbala Hospital (Other Government); Medical Centre Hungarian Defence Forces (Unknown); Hospital of Komló (Unknown); St. Pantaleon Hospital in Dunaújváros (Unknown)
Responsible Party: Sponsor
Other Study IDs: TBEP-2110/01 (2021 V2); OGYÉI/74-1/2022 (Registry Identifier: National Institute of Pharmacy and Nutrition); IV/657- 3 /2022/EKU (Registry Identifier: Medical Research Council)
Record Dates: First submitted 2022-06-27; First posted 2022-07-06 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Asthma; COPD
Keywords: aerosol drug delivery; drug delivery optimization; inhalation therapy; breathing patterns; lung deposition modelling
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Asthma patients: Patients with proven record of asthma disease.
  Interventions: Device: Emptied dry powder inhalers (DPI) used in routine asthma and COPD therapy
- COPD patients: Patients with proven record of COPD disease.
  Interventions: Device: Emptied dry powder inhalers (DPI) used in routine asthma and COPD therapy

INTERVENTIONS:
Device: Emptied dry powder inhalers (DPI) used in routine asthma and COPD therapy — The DPI inhaler devices are empty, without any active ingredient or/and carrier substances. Patients are not inhaling drug doses because of the study. They are inhaling only the type and quantity of aerosol drugs that they would inhale because of their treatment. The study does not influences the undergoing treatment by medication in any way.

SUMMARY:
This study aims to simulate the deposition of aerosol drugs within the airways of asthma and COPD patients based on realistic breathing patterns measured at different pulmonology centers.

Further goal of the study is to find correlations between the amount of drug depositing in the lungs and the measured breathing parameters, as well as disease status and demographic data. The results of the study will be part of a major objective targeting the optimization and personalization of aerosol drug therapy.

DETAILED DESCRIPTION:
The inhalation of aerosol drugs is a key element of current asthma and COPD treatment. The efficiency of the therapy is highly influenced by the dose depositing in the lungs. However, the amount of drug depositing in the lung is a result of complex drug particle-inhaler-patient interaction, thus it is inhaler-, drug- and patient-specific. Assuming that the airflow dependent aerodynamic characteristics of the drugs are known, the lung dose depends on the patient's breathing parameters during the inhalation of drug through the inhaler. In this study the inhalation parameters of asthmatic and COPD patients are measured and lung deposition assessed by a validated numerical lung deposition model. Effects of different breathing parameters (inhalation time, inhaled volume, average flow rate, peak flow rate, time until peak flow rate is reached, breath-hold time) as well as patient demographic data, disease type and disease severity on the lung dose are studied. The correlations are analysed for asthma and COPD groups separately.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed obstructive lung disease (asthma or COPD)
* proper usage of inhalation tool after being educated
* availability of whole body plethysmography measurement data from the last 6 months or the possibility to perform them before the start of the study
* subject under outpatient/inpatient therapy
* capable of acting and cooperating

Exclusion Criteria:

* the patient doesn't align with any of the criteria mentioned above
* the patient is incapable of filling out the questionnaire/questionnaires' parts that are accorded to him/her
* the patient doesn't agree to have data collected of him/her
* diagnosed heavy, not treated chronic illness
* not properly carried out /not evaluable lung function (spirometry) examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We are recruiting participants for our test from different levels of healthcare servicing (university centre, regional institute, county hospital, panel clinic) aiming to minimize centre specific effects.
Sampling Method: Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Lung deposition fraction | July 1, 2023 - June 30, 2025
  Lung deposition fraction is the ratio of the drug dose depositing in the lungs to the dose available in the device. Lung dose will be evaluated by means of computer modelling based on input data (breathing parameters) measured in this study.

SECONDARY OUTCOMES:
Inhalation time | August 1, 2022 - June 30, 2023
  Inhalation time is measured while patients inhale through the empty inhalers mimicking the inhalation of aerosol drug. It expresses the duration of the inhalation in seconds.
Peak inhalation flow | August 1, 2022 - June 30, 2023
  Peak inhalation flow is measured while patients inhale through the empty inhalers mimicking the inhalation of aerosol drug. It expresses the maximum value of the flow rate expressed in Liter/min.
Inhaled volume | August 1, 2022 - June 30, 2023
  Inhaled volume is measured while patients inhale through the empty inhalers mimicking the inhalation of aerosol drug. It expresses the quantity of inhaled air expressed in Liter.
Ramp-up time | August 1, 2022 - June 30, 2023
  Ramp-up time is determined from the inhalation curve measured while patients inhale through the empty inhalers mimicking the inhalation of aerosol drug. It expresses the time duration from the beginning of inhalation to the moment when the inhalation flow rate reaches its maximum value.
Breath-hold time | August 1, 2022 - June 30, 2023
  Breath-hold time is measured by the investigator and expresses the duration in seconds from the end of inhalation through the device until the beginning of exhalation.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Galffy, PhD, Study Director — Pest County Pulmonology Hospital
Locations (3):
- Hungary (3):
  - University of Debrecen, Debrecen
  - St. Borbala Hospital, Tatabánya
  - Pest County Pulmonology Hospital, Törökbálint

IPD SHARING:
Plan to Share IPD: Yes
The data sharing plan contains statements on the availability of individual participant data (including data dictionaries), information on what data in particular will be shared, what other documents will be available, when will data be available, with whom, for what type of analyses. In addition, the plan specifies the mechanism the data are be made available.
  According to the plan those IPD will be available that underlie the results published in research article(s) will be shared after deidentification.
  The frame of IPD sharing is defined below:
Supporting Information: Study Protocol
Time Frame: Between months 9 and 36 after the publication of article(s).
Access Criteria: IPD (individual patient data) will be shared with investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  IPD will be shared to achieve aims in the approved proposal. Proposal may be submitted to farkasar@gmail.com.
URL: https://data.mendeley.com

REFERENCES:
- [Background] Borgstrom L, Derom E, Stahl E, Wahlin-Boll E, Pauwels R. The inhalation device influences lung deposition and bronchodilating effect of terbutaline. Am J Respir Crit Care Med. 1996 May;153(5):1636-40. doi: 10.1164/ajrccm.153.5.8630614.
- [Background] Borghardt JM, Kloft C, Sharma A. Inhaled Therapy in Respiratory Disease: The Complex Interplay of Pulmonary Kinetic Processes. Can Respir J. 2018 Jun 19;2018:2732017. doi: 10.1155/2018/2732017. eCollection 2018. PMID 30018677
- [Background] Busse WW, Brazinsky S, Jacobson K, Stricker W, Schmitt K, Vanden Burgt J, Donnell D, Hannon S, Colice GL. Efficacy response of inhaled beclomethasone dipropionate in asthma is proportional to dose and is improved by formulation with a new propellant. J Allergy Clin Immunol. 1999 Dec;104(6):1215-22. doi: 10.1016/s0091-6749(99)70016-3. PMID 10589004
- [Background] Buttini F, Brambilla G, Copelli D, Sisti V, Balducci AG, Bettini R, Pasquali I. Effect of Flow Rate on In Vitro Aerodynamic Performance of NEXThaler((R)) in Comparison with Diskus((R)) and Turbohaler((R)) Dry Powder Inhalers. J Aerosol Med Pulm Drug Deliv. 2016 Apr;29(2):167-78. doi: 10.1089/jamp.2015.1220. Epub 2015 Sep 10. PMID 26355743
- [Background] Corradi M, Chrystyn H, Cosio BG, Pirozynski M, Loukides S, Louis R, Spinola M, Usmani OS. NEXThaler, an innovative dry powder inhaler delivering an extrafine fixed combination of beclometasone and formoterol to treat large and small airways in asthma. Expert Opin Drug Deliv. 2014 Sep;11(9):1497-506. doi: 10.1517/17425247.2014.928282. Epub 2014 Jun 12. PMID 24921434
- [Background] de Boer AH, Gjaltema D, Hagedoorn P, Frijlink HW. Can 'extrafine' dry powder aerosols improve lung deposition? Eur J Pharm Biopharm. 2015 Oct;96:143-51. doi: 10.1016/j.ejpb.2015.07.016. Epub 2015 Jul 26. PMID 26220014
- [Background] Horvath A, Farkas A, Szipocs A, Tomisa G, Szalai Z, Galffy G. Numerical simulation of the effect of inhalation parameters, gender, age and disease severity on the lung deposition of dry powder aerosol drugs emitted by Turbuhaler(R), Breezhaler(R) and Genuair(R) in COPD patients. Eur J Pharm Sci. 2020 Nov 1;154:105508. doi: 10.1016/j.ejps.2020.105508. Epub 2020 Aug 21. PMID 32836137
- [Background] Horvath A, Balashazy I, Tomisa G, Farkas A. Significance of breath-hold time in dry powder aerosol drug therapy of COPD patients. Eur J Pharm Sci. 2017 Jun 15;104:145-149. doi: 10.1016/j.ejps.2017.03.047. Epub 2017 Apr 4. PMID 28389274
- [Background] Jokay A, Farkas A, Furi P, Horvath A, Tomisa G, Balashazy I. Computer modeling of airway deposition distribution of Foster((R)) NEXThaler((R)) and Seretide((R)) Diskus((R)) dry powder combination drugs. Eur J Pharm Sci. 2016 Jun 10;88:210-8. doi: 10.1016/j.ejps.2016.03.008. Epub 2016 Mar 11. PMID 26976481
- [Background] Virchow JC, Poli G, Herpich C, Kietzig C, Ehlich H, Braeutigam D, Sommerer K, Haussermann S, Mariotti F. Lung Deposition of the Dry Powder Fixed Combination Beclometasone Dipropionate Plus Formoterol Fumarate Using NEXThaler(R) Device in Healthy Subjects, Asthmatic Patients, and COPD Patients. J Aerosol Med Pulm Drug Deliv. 2018 Oct;31(5):269-280. doi: 10.1089/jamp.2016.1359. Epub 2018 Jul 10. PMID 29989511
- [Background] Prime D, de Backer W, Hamilton M, Cahn A, Preece A, Kelleher D, Baines A, Moore A, Brealey N, Moynihan J. Effect of Disease Severity in Asthma and Chronic Obstructive Pulmonary Disease on Inhaler-Specific Inhalation Profiles Through the ELLIPTA(R) Dry Powder Inhaler. J Aerosol Med Pulm Drug Deliv. 2015 Dec;28(6):486-97. doi: 10.1089/jamp.2015.1224. Epub 2015 Sep 15. PMID 26372467
- [Background] Hamilton M, Leggett R, Pang C, Charles S, Gillett B, Prime D. In Vitro Dosing Performance of the ELLIPTA(R) Dry Powder Inhaler Using Asthma and COPD Patient Inhalation Profiles Replicated with the Electronic Lung (eLung). J Aerosol Med Pulm Drug Deliv. 2015 Dec;28(6):498-506. doi: 10.1089/jamp.2015.1225. Epub 2015 Sep 15. PMID 26372465
- See also: Global Initiative for asthma (GINA) — https://ginasthma.org
- See also: Global Initiative for Chronic Obstructive Lung Disease (GOLD) — https://goldcopd.org

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT05445349/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT05445349/ICF_001.pdf